CLINICAL TRIAL: NCT01763671
Title: Phase III Study Comparing the Efficacy of Paclitaxel-bevacizumab With Docetaxel in 2nd or 3rd Line of Treatment of Non Squamous Non Small Cells Lung Cancer
Brief Title: Paclitaxel-bevacizumab in Advanced Lung Cancer
Acronym: Ultimate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-1103
Record Dates: First submitted 2013-01-07; First posted 2013-01-09 (Estimated); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Non-squamous Non-small Cell Lung Cancer
Keywords: Lung cancer; Paclitaxel bevacizumab; IFCT
MeSH Terms: conditions — Lung Neoplasms | interventions — Docetaxel; Paclitaxel; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Docetaxel (Active Comparator)
  Interventions: Drug: Docetaxel
- Paclitaxel - Bevacizumab (Experimental)
  Interventions: Drug: Paclitaxel; Drug: Bevacizumab

INTERVENTIONS:
Drug: Docetaxel — 75 mg/m² IV on day one of 21 days cycle Number of Cycles: until progression or unacceptable toxicity develops.
  Arms: Docetaxel
Drug: Paclitaxel — 90 mg/m² IV on day 1, 8 and 15 of 28 days cycle Number of Cycles: until progression or unacceptable toxicity develops.
  Arms: Paclitaxel - Bevacizumab
Drug: Bevacizumab — 10 mg/kg IV on day 1 and 15 of 28 days cycle Number of Cycles: until progression or unacceptable toxicity develops.
  Arms: Paclitaxel - Bevacizumab

SUMMARY:
The study objective is to evaluate the efficacy of paclitaxel-bevacizumab comparing to docetaxel.

Docetaxel is a standard treatment of 2nd or 3rd line in lung cancer. It was validated by numerous clinical trials but sometimes toxicities are difficult to manage.

Bevacizumab is an antiangiogenic treatment which was validated by numerous clinical trials in association with platinum in first ligne. Different clinical and preclinical data suggest that there could exist a synergy between paclitaxel and bevacizumab. This association is already used in metastatic breast cancer, it permits almost to double the response rate and progression free survival. In lung cancer, the association was evaluated by two retrospective studies which demonstrated a benefit with a favourable safety profile.

ELIGIBILITY:
Inclusion Criteria:

* 2nd or 3rd line of non squamous non small cell lung cancer of stage III or IV
* Document progression at the time of the inclusion. At least, one previous chemotherapy line with platinum. Patient who had previous treatment with bevacizumab can be included.
* Patient with active mutation of EGFR must have had on line of chemotherapy with platinum and one with Tyrosine kinase inhibitor of EGFR.
* Patient with ALK rearrangement must have had at least one line of chemotherapy with platinum and one with crizotinib.

Exclusion Criteria:

* Mixed cancer small cells and non small cells or squamous lung cancer.
* Central nervous system symptomatic metastasis or requiring immediate cerebral radiotherapy
* patient who have had previous treatment with taxane (docetaxel, paclitaxel). Peri-operatory chemotherapy or chemoradiotherapy with taxane allowed if stopped more than 6 months before.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2013-05; Primary Completion 2015-12 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Progression free survival | about 4 months
  Time between inclusion and progression

SECONDARY OUTCOMES:
Response Rate | At 8 weeks
Overall survival | about 8 months
  Time between inclusion and death

CONTACTS AND LOCATIONS:
Overall Officials: Alexis CORTOT, MD, Principal Investigator — CHRU LILLE; Benjamin BESSE, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (55):
- France (55):
  - Amiens - CHU, Amiens
  - Centre Hospitalier, Annemasse
  - Hôpital Privé d'Antony, Antony
  - Avignon - Institut Sainte-Catherine, Avignon
  - CH de la Côte Basque, Bayonne
  - Béziers - CH, Béziers
  - Bordeaux - Polyclinique Nord, Bordeaux
  - Caen - Centre François Baclesse, Caen
  - Caen - CHU Côte de Nacre, Caen
  - Castelnau Le Lez - Clinique, Castelnau
  - CH de Chartres Hôpital Louis Pasteur, Chartres
  - Chauny - CH, Chauny
  - CH, Cholet
  - Hôpital Percy-Armées - Pneumologie, Clamart
  - Hôpitral Gabriel Montpied - Pneumologie, Clermont-Ferrand
  - CH, Colmar
  - CH Compiègne - Pneumologie, Compiègne
  - CHI Créteil, Créteil
  - CHRU Grenoble, Grenoble
  - Harfleur - Clinique du Petit Colmoulins, Harfleur
  - CH Région Saint-Omer, Helfaut
  - Le Mans - Centre Hospitalier, Le Mans
  - CHU (Hôpital Calmette) - Pneumologie, Lille
  - CH de Longjumeau, Longjumeau
  - Lorient - CHBS, Lorient
  - Lyon - Hôpital Jean Mermoz, Lyon
  - Lyon - Hôpital Louis Pradel (Pneumologie), Lyon
  - Mantes La Jolie - CH, Mantes-la-Jolie
  - Marseille - Hôpital Sainte Marguerite, Marseille
  - Maubeuge - Polyclinique du Parc, Maubeuge
  - CH de Macon, Mâcon
  - CH Montélimar, Montélimar
  - Mulhouse - CH, Mulhouse
  - Nantes - Centre René Gauducheau, Nantes
  - CHR d'Orléans La Source, Orléans
  - Paris - Saint Louis, Paris
  - Hopital Tenon - Pneumologie, Paris
  - HIA Val-de-Grâce, Paris
  - Hôpital Bichat - Claude - Bernard, Paris
  - Paris - Pitié-salpêtrière, Paris
  - Pau - CH, Pau
  - Lyon Sud, Pierre-Bénite
  - Rouen - CHU, Rouen
  - CHU Saint-Etienne Pneumologie, Saint-Etienne
  - Saint Quentin - CH, Saint-Quentin
  - Strasbourg - NHC, Strasbourg
  - Suresnes - Hopital Foch, Suresnes
  - Thonon les bains - CH, Thonon-les-Bains
  - Toulon - CHI, Toulon
  - Toulon - HIA, Toulon
  - Toulouse - CHU Larrey, Toulouse
  - Tours - CHU, Tours
  - Valenciennes - Clinique, Valenciennes
  - CH de Villefranche - Pneumologie, Villefranche
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Cortot AB, Audigier-Valette C, Molinier O, Le Moulec S, Barlesi F, Zalcman G, Dumont P, Pouessel D, Poulet C, Fontaine-Delaruelle C, Hiret S, Dixmier A, Renault PA, Becht C, Raffy O, Dayen C, Mazieres J, Pichon E, Langlais A, Morin F, Moro-Sibilot D, Besse B. Weekly paclitaxel plus bevacizumab versus docetaxel as second- or third-line treatment in advanced non-squamous non-small-cell lung cancer: Results of the IFCT-1103 ULTIMATE study. Eur J Cancer. 2020 May;131:27-36. doi: 10.1016/j.ejca.2020.02.022. Epub 2020 Apr 8. PMID 32276179
- See also: Official IFCT website — https://www.ifct.fr/etudes-cliniques/420-ifct-1103